CLINICAL TRIAL: NCT06557148
Title: 18F-Fluoroestradiol (FES) Positron Emission Tomography for the Detection and Treatment Response Monitoring in Patients With Metastatic Lobular Breast Carcinoma
Brief Title: A Study Comparing Cancer Imaging Approaches in People With Lobular Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 24-134
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Lobular Breast Carcinoma; Breast Carcinoma; Metastatic Breast Cancer; Metastatic Lobular Breast Carcinoma; Metastatic Breast Carcinoma
Keywords: breast cancer; lobular breast cancer; lobular breast carcinoma; breast carcinoma; metastatic breast cancer; metastatic lobular breast cancer; metastatic lobular breast carcinoma; metastatic breast carcinoma; 24-134; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Lobular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biopsy-proven ER+ Metastatic Invasive Lobular Carcinoma/ILC: Participants will have biopsy-proven metastatic ILC, confirmed ER+ breast cancer
  Interventions: Diagnostic Test: 18F-Fluoroestradiol PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-Fluoroestradiol PET/CT — Scanned at baseline and again posttreatment within 2 weeks of the restaging FDG PET/CT
  Other Names: FES PET/CT

SUMMARY:
The purpose of this study to compare two types of cancer imaging scans to see which is better at detecting and monitoring metastatic ILC. This study will compare PET/CT (positron emission tomography/computed tomography) scans using the radiotracer fluorine 18 (18F)-fluoroestradiol (FES) with a standard imaging approach for detecting and monitoring ILC, PET/CT scans using the radiotracer 18F-fluorodeoxyglucose (FDG). These scans will be referred to as FES PET/CT scans and FDG PET/CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 18 years old
* Biopsy-proven metastatic ILC
* Confirmed ER+ breast cancer from either primary tumor or metastatic biopsy (ER receptor percent staining ≥ 10% of tumor cells by IHC)
* HER2-negative per ASCO/CAP
* ECOG Performance Status Score of 0, 1 or 2.
* Patient can have received up to 2 lines of therapy in the metastatic setting
* Life expectancy of at least 12 months

Exclusion Criteria:

* Low ER expression defined as ER <10% of tumor cells by IHC
* Patients who have been on adjuvant ER-blocking endocrine therapy with SERM or SERD without an 8- and 24-weeks washout, respectively. (The use of aromatase inhibitors or ovarian suppression is permitted given that they do not block estrogen receptors).
* Pregnancy or lactation or parturient or nursing mother
* Patient presents with any other clinically active, serious, life-threatening disease, medical, or psychiatric condition, and/or who has a life expectancy of <12 months, or for whom study participation may compromise their management; and/or a patient who the investigator judges to be unsuitable for participation in the study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from breast medical oncology clinics, with a concerted effort to recruit a diverse group of patients. Recruitment will be led by Co-PI Komal Jhaveri, MD, Assistant Attending, Breast Medicine Service. Eligible patients will be approached to enroll in the protocol and provide written informed consent. Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at MSK. If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-08-13 (Estimated); Study Completion 2027-08-13 (Estimated)

PRIMARY OUTCOMES:
Comparison of FES PET/CT in Metastatic Invasive Lobular Carcinoma/ILC to standard-of-care (SOC) imaging with FDG PET/CT at baseline | 1 year
  Disease detection by 18F-FES and 18F-FDG PET/CT images at baseline will be directly compared

CONTACTS AND LOCATIONS:
Overall Officials: Somali Gavane, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org